CLINICAL TRIAL: NCT03185351
Title: Perineural Versus Intravenous Midazolam in Patients Undergoing Forearm Orthopedic Surgeries Using Supraclavicular Brachial Plexus Block
Brief Title: Midazolam in Supraclavicular Brachial Plexus Block
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, RAGAA AHMED HERDAN, Lecturer of Anesthesia and Intensive Care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: brachial plexus block
Record Dates: First submitted 2017-05-21; First posted 2017-06-14 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Forearm Surgeries
Keywords: midazolam; brachial plexus block
MeSH Terms: interventions — Bupivacaine; Midazolam

STUDY DESIGN:
Intervention Model Description: * Group A: patients will receive 20 ml of 0.5% bupivacaine + 5 ml normal saline (0.9%) using supraclavicular BPB.
  * Group B: patients will receive 20 ml of 0.5% bupivacaine + midazolam 0.03 mg/kg dissolved in 5 ml normal saline (0.9%) using supraclavicular BPB.
  * Group C: patients will receive 20 ml of 0.5% bupivacaine + 5 ml normal saline (0.9%) using supraclavicular BPB + 0.03 mg/kg of midazolam by I.V. route at the same time of the block.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BUPIVACAINE (Active Comparator): patients will receive 20 ml of 0.5% bupivacaine + 5 ml normal saline (0.9%) using supraclavicular BPB.
  .
  Interventions: Drug: Bupivacaine
- BUPIVACAINE and midazolam (Active Comparator): patients will receive 20 ml of 0.5% bupivacaine + midazolam 0.03 mg/kg dissolved in 5 ml normal saline (0.9%) using supraclavicular BPB.
  Interventions: Drug: Bupivacaine; Drug: Midazolam
- BUPIVACAINE and i.v midazolam (Active Comparator): patients will receive 20 ml of 0.5% bupivacaine + 5 ml normal saline (0.9%) using supraclavicular BPB + 0.03 mg/kg of midazolam by I.V. route at the same time of the block
  Interventions: Drug: Bupivacaine; Drug: Midazolam

INTERVENTIONS:
Drug: Bupivacaine — 20 ml of 0.5% bupivacaine using supraclavicular BPB.
Drug: Midazolam — midazolam 0.03 mg/kg dissolved in 5 ml normal saline (0.9%) using supraclavicular BPB
  Arms: BUPIVACAINE and midazolam
Drug: Midazolam — 0.03 mg/kg of midazolam by I.V. route
  Arms: BUPIVACAINE and i.v midazolam

SUMMARY:
An effective brachial plexus block (BPB) provides a useful alternative to general anesthesia for upper arm surgery producing complete muscular relaxation. It provides surgical anesthesia in upper extremity surgery, post-operative analgesia and chronic pain management. In addition to surgical procedure on conscious patients and early eating after the procedure make regional anesthesia more attractive.

Brachial plexus block also maintains stable intraoperative hemodynamic and associated sympathetic block. The sympathetic block decreases postoperative pain, vasospasm and edema. The nerve of brachial plexus may be blocked anywhere along its course. The approach for blocking brachial plexus nerve is interscalene, supraclavicular, infraclavicular and axillary approach.

Supraclavicular approach for blockade of the brachial plexus is the most commonly used approach in providing surgical anesthesia. In recent years, the technique has gained importance as regional anesthetic technique for surgical, diagnostic and therapeutic purposes in interventional pain management. It includes blocking of the brachial plexus where it is most compactly arranged, with fewer requirements of the anesthetic solution and rapid onset of action. Supraclavicular nerve block is technically easy to perform because of reliable and fixed landmark but association of pneumothorax is a profound complication.

The extent of blockade following injection into the sheath surrounding the brachial plexus may depend on the volume and concentration of local anesthetic (LA) used. Because of bupivacaine long duration of action, it is used most frequently among local anesthetics for BPB.

Inevitably, the effects of single-injection BPB dissipate after several hours unmasking the moderate-to-severe pain of the surgical insult. Efforts to prolong BPB duration by increasing LA dose are limited by their narrow therapeutic window and indeed may not be effective as recent studies have demonstrated equivalent analgesic duration with volumes as low as 5 ml.

Midazolam is known to produce antinociception and potentiate the effect of LA when given in neuraxial block. It produces this effect by its action on Gamma Aminobutyric Acid-A (GABA-A) receptors and also on the peripheral nerves which contain these receptors.

Several studies showed midazolam to be effective when used in intrathecal, epidural and caudal blocks and now recently midazolam with bupivacaine has been found to improve analgesic characteristics in peripheral blocks compared to bupivacaine alone. Due to the high blood concentration of benzodiazepine through conventional routes and profound sedation, proper assessment of analgesic effect was difficult to obtain. With the advent of the less toxic water soluble benzodiazepine (midazolam), it became possible to use it directly over the nerve tissues.

DETAILED DESCRIPTION:
The day prior to surgery, all patients will undergo pre-anesthetic checkup including detailed history, thorough general, physical, systemic examination and weight of the patient. All patients will be kept nil by mouth for at least 6 hours.

* Written consent, coagulation profile, intravenous line, emergency resuscitation equipments including airway devices, advanced cardiac life support drugs for LA toxicity will be available.
* Patients will be monitored using standard monitoring (ECG, non-invasive blood pressure and pulsoximetry)
* All patients will be lightly sedated with 1 mg midazolam I.V. SonoAce 6 ultrasound machine with high frequency linear probe will be used in our study.

Palpation of the subclavian artery in the supraclvicular fossa, just lateral to the sternocledomastoid and above the clavicle (landmark located one finger or 1 cm above the clavicle at the junction of inner 2/3 and outer 1/3 of clavicle).

Position to perform supraclavicular BPB; the anesthetist will stand behind the patient's head, with the ultrasound machine on the side being blocked. The head of the bed is slightly raised to allow the shoulder to drop somewhat the patient's head will be turned to the opposite side, resting directly on the table without a pillow, the hand holding the probe will rest against the patient's jaw, the probe is placed in the supraclavicular fossa in a coronal oblique plane, the needle will be inserted from the lateral side, The pulsating hypoechoic supraclavicular artery is identified, lying above the hyperechoic first rib, the probe is then angled until both the first rib and the pleura are also seen simultaneously, The nerve structures (trunks or divisions) are usually visualized as a collection of hypoechoic round structures (a bunch of grapes) lying superior and postero-lateral to the subclavian artery. A 3 cm long 22 G needle with 10 cc syringe filled with respective LA agent will be inserted directing downward, forward and medially at the angle of 20° to the skin till the parasthesia elicited in the hand or the 1st rib hit, then the needle will be fixed at that point. After the negative aspiration respective agents will be given. A gentle massage over the area will be done with an idea of uniform spread. All brachial plexus injections will be administered slowly with repeated aspiration to prevent or detect early intravascular injection. The end of the injection will be considered time 0.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II physical status patients.
* Age between 18 and 50 years.
* Patients planned for unilateral orthopedic forearm surgeries.

Exclusion Criteria:

* Patient refusal
* Any contraindication to regional block (i.e. coagulopathy, infection at the needle insertion site, contralateral pneumothorax or diaphragmatic paralysis)
* Bilateral limb surgery
* Pregnancy
* BMI >35
* Preexisting neuropathy involving the surgical limb
* Patients with any known contraindication to study medications
* History of a major psychiatric disorder.
* Chronic pain syndrome.
* History of substance abuse.
* Current opioid use.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Numerical rating pain scale graded from 0 to 10 | 24 hours
  postoperative analgesic efficacy of ultrasound guided supraclavicular BPB

SECONDARY OUTCOMES:
Motor blockade | 24 hours
  Modified Bromage Score
Sedation Score | 24 hours
  (Awake and alert -1, Sedated and responding to verbal command-2, Sedated and responding to mild stimulus-3, Sedated and responding to moderate to severe physical stimulus-4).

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided